CLINICAL TRIAL: NCT06668103
Title: A Phase 2, Open-Label Study to Evaluate the Efficacy and Safety of ABSK043 Combined With Firmonertinib in Patients With EGFR Mutated Locally Advanced or Metastatic Non-small Cell Lung Cancer(NSCLC)
Brief Title: A Phase 2 Clinical Study of Combination Therapy With ABSK043 and Firmonertinib
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Abbisko Therapeutics Co, Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ABSK043-202
Record Dates: First submitted 2024-10-30; First posted 2024-10-31 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-10

CONDITIONS: Non-Small Cell Lung Cancer With EGFR Mutation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ABSK043 in combination with Firmonertinib (Experimental): This is an open-label phase 2 study with an escalation part and an expansion part.
  * Escalation part: Previously treated patients with EGFR Mutated NSCLC will be enrolled.
    * Dose escalation cohort: up to 12 patients;
    * Dose confirmation cohort: at least 3 patients, and up to 12 patients.
  * Expansion part:
    * Dose expansion cohort: up to 30 treatment-naïve patients with EGFR Mutated NSCLC are expected to be enrolled.
  Interventions: Drug: ABSK043 in combination with Firmonertinib

INTERVENTIONS:
Drug: ABSK043 in combination with Firmonertinib — Two potential dose levels ：400 mg twice daily （BID） and 800 mg BID) of ABSK043 are prespecified and firmonertinib will be administered orally at a fixed dose of 80 mg once daily (QD).
  Patients in dose escalation cohort will receive the ABSK043, 400 mg BID and firmonertinib 80 mg QD as the starting dose for the combination therapy.
  Patients in dose confirmation cohort and dose expansion cohort will receive the recommended dose in dose escalation cohort and be evaluated for safety and preliminary anti-tumor activity of the combination therapy.
  After Cycle 1, patients will continue to receive combination therapy every 21 days until disease progression, death, loss to follow-up, withdrawal of consent, intolerable toxicity, investigator decision to discontinue treatment, or end of the study.

SUMMARY:
This is an open-label phase 2 study to evaluate the safety, tolerability and preliminary anti-tumour activity of ABSK043 in combination with Firmonertinib in patients with Epidermal Growth Factor Receptor-mutated (EGFRm+) locally advanced or metastatic NSCLC.

DETAILED DESCRIPTION:
This is a Phase II, open-label, multicentre study of ABSK043 administered orally in combination with Firmonertinib to patients with EGFRm+ advanced NSCLC. The study has been designed to allow an investigation of the optimal combination dose and schedule whilst ensuring the safety of patients with intensive safety monitoring. There are two main parts to this study; Part A, dose escalation and Parts B Dose expansion. The expansion part will evaluate the efficacy of ABSK043 in combination with Firmonertinib as first-line treatment for locally advanced or metastatic NSCLC patients with EGFR-mutated at the one or more recommended dose.

Dose escalation:

• Post-line: Patients with locally advanced or metastatic NSCLC with an EGFR exon 19 deletion or L858R mutation with tumor progression after treatment with systemic treatment

Dose Expansion:

• First-Line: Patients with locally advanced or metastatic NSCLC with an EGFR exon 19 deletion or L858R mutation, and without prior systemic therapy for advanced or metastatic disease.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically documented locally advanced or metastatic NSCLC
2. At least 1 measurable lesion as assessed by Investigator as per Response Evaluation Criteria in Solid Tumors (RECIST v1.1)
3. Inclusion Criteria Specific to Dose Escalation cohort and Dose Confirmation Cohort：Must has disease progression following treatment with EGFR-TKI in the locally advanced or metastatic setting for locally advanced or metastatic disease Documentation of PDL1 expression positive (TPS/TC≥1%)detected from tumor tissue Inclusion Criteria Specific to Dose expansion Cohort： Must not have received any other prior systemic cancer therapies in the locally advanced/metastatic setting PDL1 expression positive (TPS/TC≥1%) as assessed by central laboratory from tumor tissue
4. Adequate bone marrow reserve and organ function based on local laboratory data .
5. Documented genetic testing reports confirmed the presence of EGFR L858R or EGFR exon 19 del mutations in tumor or plasma ctDNA.

Exclusion Criteria:

1. 1. Histological or cytological examinations suggest that NSCLC squamous cells is the predominant histology, or contains small cell lung cancer, neuroendocrine carcinoma, etc.
2. Has a history of interstitial lung disease (ILD)/pneumonitis or active ILD
3. Has spinal cord compression or clinically active central nervous system metastases, defined as symptomatic, or requiring therapy with corticosteroids or anticonvulsants to control associated symptoms. Participants with clinically inactive brain metastases may be included in the study
4. Has unresolved toxicities from previous anticancer therapy, defined as toxicities (other than alopecia) not yet resolved to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0, Grade ≤1 or baseline.
5. Is receiving chronic systemic corticosteroids dosed at >10 mg prednisone or equivalent anti-inflammatory activity or any form of immunosuppressive therapy.
6. Uncontrolled or significant cardiovascular disease
7. Has a known human immunodeficiency virus (HIV) infection that is not well controlled.
8. Any evidence of severe or uncontrolled diseases or other factors which in the Investigator's opinion makes it undesirable for the patients to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2024-11-25 (Actual); Primary Completion 2027-12-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of DLT | At the end of Cycle 1 (each cycle is 21 days)
  Dose-limiting toxicities
AEs | From the time the patient signs the informed consent form throughout the study and up to 90 days after the last dose of ABSK043 or 30 days after the last dose of furmonertinib mesylate, whichever occurs first, up to 30 months.
  Adverse events
SAEs | From the time patients sign the informed consent form throughout the study and up to 90 days after the last dose of ABSK043 or 30 days after the last dose of furmonertinib mesylate, whichever occurs first, up to 30 months.
  Serious adverse events (SAEs)
AESIs | From the time patients sign the informed consent form throughout the study and up to 90 days after the last dose of ABSK043 or 30 days after the last dose of furmonertinib mesylate, whichever occurs first, up to 30 months.
  Adverse events of special interest (AESIs)
PFS rate at 12 month | From the time patients receive the first dose of study drug to 12 months，assessed up to 30 months.
  Progression-free survival at 12 month

SECONDARY OUTCOMES:
Cmax | From the date of enrolment #Cycle1 Day1# to #Cycle7#, and for patients who discontinue treatment before cycle 7 (C7), PK sampling will be performed at the EOT visit and assessed up to 10 months.
  Maximum observed concentration
AUC | From the date of enrolment #Cycle1 Day1# to #Cycle7#, and for patients who discontinue treatment before cycle 7 (C7), PK sampling will be performed at the EOT visit and assessed up to 10 months.
  area under the concentration-time curve area under the concentration-time curve area under the concentration-time curve
t1/2 | From the date of enrolment #Cycle1 Day1# to #Cycle7#, and for patients who discontinue treatment before cycle 7 (C7), PK sampling will be performed at the EOT visit and assessed up to 10 months.
  elimination half-life
Vz/F | From the date of enrolment #Cycle1 Day1# to #Cycle7#, and for patients who discontinue treatment before cycle 7 (C7), PK sampling will be performed at the EOT visit and assessed up to 10 months.
  apparent volume of distribution
CL/F | From the date of enrolment #Cycle1 Day1# to #Cycle7#, and for patients who discontinue treatment before cycle 7 (C7), PK sampling will be performed at the EOT visit and assessed up to 10 months.
  apparent oral clearance
Cmax,ss | From the date of enrolment #Cycle1 Day1# to #Cycle7#, and for patients who discontinue treatment before cycle 7 (C7), PK sampling will be performed at the EOT visit and assessed up to 10 months.
  maximum observed concentration after multiple doses
Cmin,ss | From the date of enrolment #Cycle1 Day1# to #Cycle7#, and for patients who discontinue treatment before cycle 7 (C7), PK sampling will be performed at the EOT visit and assessed up to 10 months.
  minimum observed concentration after multiple doses
AUCtau,ss | From the date of enrolment #Cycle1 Day1# to #Cycle7#, and for patients who discontinue treatment before cycle 7 (C7), PK sampling will be performed at the EOT visit and assessed up to 10 months.
  area under the concentration-time curve after multiple doses
AR | From the date of enrolment #Cycle1 Day1# to #Cycle7#, and for patients who discontinue treatment before cycle 7 (C7), PK sampling will be performed at the EOT visit and assessed up to 10 months.
  accumulation ratio
tmax | From the date of enrolment #Cycle1 Day1# to #Cycle7#, and for patients who discontinue treatment before cycle 7 (C7), PK sampling will be performed at the EOT visit and assessed up to 10 months.
  time to maximum observed concentration
ORR | From date of enrolment#Cycle1 Day1# until disease progression, death, loss to follow-up, withdrawal of consent, intolerable toxicity, investigator's decision to discontinue treatment, or end of study, whichever comes first, assessed up to 30 months.
  Objective response rate
DOR | From date of enrolment#Cycle1 Day1# until disease progression, death, loss to follow-up, withdrawal of consent, intolerable toxicity, investigator's decision to discontinue treatment, or end of study, whichever comes first, assessed up to 30 months.
  Duration of response
PFS | From date of enrolment#Cycle1 Day1# until disease progression, death, loss to follow-up, withdrawal of consent, intolerable toxicity, investigator's decision to discontinue treatment, or end of study, whichever comes first, assessed up to 30 months.
  Progression-free survival
DCR | From date of enrollment#Cycle1 Day1# until disease progression, death, loss to follow-up, withdrawal of consent, intolerable toxicity, investigator decision to discontinue treatment, or end of the study, whichever comes first，assessed up to 30 months.
  Disease control rate
OS | From date of enrolment#Cycle1 Day1# until disease progression, death, loss to follow-up, withdrawal of consent, intolerable toxicity, investigator's decision to discontinue treatment, or end of study, whichever comes first, assessed up to 30 months.
  Overall survival
TTP | From date of enrolment #Cycle1 Day1# until disease progression, assessed up to 30 months.
  Time to progression

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - Hanhui Cancer Hospital, Hefei, Anhui
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Union Hospital Tongji Medical College Huzhong University of Science and Techology, Wuhan, Hubei
  - Jilin Cancer Hospital, Changchun, Jilin
  - Shanghai Chest Hospital, Shanghai, Shanghai Municipality